CLINICAL TRIAL: NCT06699888
Title: Effect of Cervicothoracic Junction Manipulation on Craniovertebral Angle and Proprioception in Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Riphah IU Samiyah Asghar
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Forward Head Posture
Keywords: Cervicothoracic Manipulation; Craniovertebral Angle; Joint position Error; Proprioception

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervicothoracic Manipulation group (Experimental): the subject will receive cervicothoracic manipulation and Chin tuck, Strengthening Shoulder Retractors, Stretching SCM, Pectoralis Stretch
  Interventions: Other: cervicothoracic manipulation group
- forward head correction exercises group (Active Comparator): this group receive Chin tuck, Strengthening Shoulder Retractors, Stretching SCM, Pectoralis Stretch
  Interventions: Other: forward head correction exercises traditional group

INTERVENTIONS:
Other: cervicothoracic manipulation group — The participant lay prone with the head firmly into the head piece Palpation of the upper cervico-thoracic segment observed the side of the restriction.
  The participants head was rotated to the contralateral side of the restriction. The practitioner's hand contacted the forehead and the other hand's thumb contacted the spinous process of the restricted side.
  A low amplitude, high velocity thrust towards the axilla was applied, on the spinous process in PA direction.
  Experimental group also received following exercises Chin tuck Strengthening Shoulder Retractors. Stretching SCM Pectoralis Stretch 3 × 10 repetitions, 3 times a week for 2 weeks
  Arms: Cervicothoracic Manipulation group
Other: forward head correction exercises traditional group — Chin tuck Strengthening Shoulder Retractors. Stretching SCM Pectoralis Stretch 3 × 10 repetitions, 3 times a week for 2 weeks.
  Arms: forward head correction exercises group

SUMMARY:
The aim of this research is to find out the effect of Cervicothoracic Junction Manipulation on neck Proprioception in individuals with Forward Head Posture. A Randomized controlled trials done at Barki Advance Physiotherapy Center. The sample size was 36. The subjects were divided in two groups, 18 subjects in control group and 16 in experimental (Cervicothoracic Manipulation) group. Study duration is of 6 months after the ethical approval. Sampling technique applied was non probability connivance sampling technique. Only 18-45 years individuals with forward head posture, craniovertebral angle less than 53° degrees and Joint position error, an average of >4.5◦ error in rotation or extension direction were included. Tools used in the study are Craniovertebral Angle (CVA) and Joint Position Error Test (JPE).

DETAILED DESCRIPTION:
FHP is greatly linked with multiple musculoskeletal conditions like head and neck dysfunction, myofascial trigger points, temporomandibular dysfunction, poor cervical mobility and functional disability of the cervical and thoracic spines. It also observed in asymptomatic individuals. Muscle spindles, especially in cervical detect muscle length changes and contribute to proprioception. Changes in neck muscles can disrupt proprioceptive function in the cervical spine. Proprioception is vital for joint function, providing stability during activities and informing posture and movement. Decreased balance and positioning errors are common in individuals with neck discomfort, emphasizing the importance of restoring proprioceptive function, particularly in Forward Head Posture (FHP) patients, for maintaining normal neck posture. Abnormalities in the head posture are absolutely harmful for the Head and neck posture. A study investigated the CV angle and joint position error in the cervical region and found a negative correlation between head posture and proprioceptive function, indicating that chronic abnormal head posture (FHP) negatively affects proprioception, body stability, and neck pain. Spinal manipulation uses high velocity and low amplitude thrusts to realign restricted vertebrae, removing restriction in facet joints, and producing mechanical, physiological, and biological effects.

Literature suggest that manipulation has beneficial effects in improving the pain and postural control in spine. The cervicothoracic (CT) junction is the transitional segment between the mobile lordotic cervical and less mobile kyphotic thoracic spines and hence a potential region for stiffness. The cervicothoracic junction, a potential stiffness region, can cause neck, headache, and upper limb pain. Improving its range of motion could reduce the need for compensatory movement, reducing cervical spine tension. According to recent systematic review, cervicothoracic junction level manual therapy in subjects with FHP better improved the muscle recruitment ability than upper-cervical level manual therapy during motor tasks. Upper thoracic spine manipulation has been shown to be more beneficial than thoracic mobilization, cervical mobilization, and standard care for FHP during performing motor task. In 2023 study conducted by Ibrahim et al. find out that FHP influenced Somatosensory Evoked Potentials and Somatosensory Processing in asymptomatic young adults and they reported 1-degree increase in the CVA measurement (indicating better posture) significantly decreased the amplitudes of all the potentials and resulted in a faster, more efficient nerve conduction time

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients with age between 18-45 years
* Participants with asymptomatic Forward head posture
* Participants having no active complain of neck pain and muscle stiffness
* Joint position error, an average of >4.5◦ error in rotation or extension directions
* For FHP patient, the Craniovertebral angle should be ≤ 53º

Exclusion Criteria:

* Previous history of neck and head trauma
* Vestibular pathologies i.e. vertigo, dizziness
* Musculoskeletal or neurological conditions that could affect Proprioception, cognitive impairment
* History of spinal and thoracic surgeries

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Craniovertebral Angle | baseline to 2 weeks
  The CV angle was measured for assessment of head posture. All subjects were instructed to stand in a self-selected comfortable upright posture. Then, the skin overlying the spinous process of the seventh cervical vertebra (C7) and tragus of the ear was marked. A lateral view digital photograph of each subject was taken. The CV angle was calculated based on the angle between a horizontal line passing through C7 and a line extending from the tragus of the ear to C7. The x-axis values for the craniovertebral angle were measured prior to movement.
Joint Position Error Test | baseline to 2 weeks
  Proprioceptive accuracy, pertaining to the sense of joint and body movement and position, was evaluated using the Joint Position Error (JPE) Test. The Cervical JPE Test measures the ability of a blindfolded patient to accurately relocate their head position back to a predetermined neutral point after cervical joint movement

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Barki Rehabilitation Center, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No